CLINICAL TRIAL: NCT07087418
Title: AI-Driven Multimodal Imaging Integration for Diagnosis and Prognostication of Digestive System Diseases
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xuehua Li, associate chief physician, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 82270693
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Digestive Diseases; Radiology; AI (Artificial Intelligence); Imaging
Keywords: Radiology; Imaging; Digestive Diseases; Artificial Intelligence
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional endoscopy group: Prognostic indicators (e.g., clinical remission rate, recurrence risk) were predicted using conventional endoscopy at baseline.
  Interventions: Diagnostic Test: Kaplan-Meier analysis with log-rank testing
- Virtual endoscopy group: Prognostic indicators were predicted using virtual endoscopy at baseline.
  Interventions: Diagnostic Test: Kaplan-Meier analysis with log-rank testing

INTERVENTIONS:
Diagnostic Test: Kaplan-Meier analysis with log-rank testing — The non-inferiority of the virtual endoscopy group will be verified by comparing the predictive performance for prognostic indicators (e.g., clinical remission rate, recurrence risk) between the two groups during follow-up.

SUMMARY:
The goal of this observational study is to to develop a noninvasive disease assessment system by leveraging artificial intelligence (AI) to comprehensively analyze multi-modal imaging features, including magnetic resonance enterography (MRE) and computed tomography enterography (CTE), for the diagnosis and prognostication of digestive diseases.

Participants will be randomly assigned to either conventional endoscopy or virtual endoscopy groups. The predictive performance of both groups for prognostic indicators, such as clinical remission rate and recurrence risk, will be compared during follow-up to verify the non-inferiority of the virtual endoscopy group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multimodal-confirmed diagnoses (clinical, imaging, endoscopic, and pathological) of:

  * Inflammatory bowel disease (IBD; Crohn's disease or ulcerative colitis)
  * Intestinal tuberculosis
  * Behçet's disease
* Availability of ≥1 technically adequate CT or MR scan with high-quality colonoscopy performed within ±1 month of imaging.

Exclusion Criteria:

* ・Suboptimal imaging quality (e.g., low-dose artifacts, metal artifacts)

  * Inadequate bowel preparation for endoscopy
  * Incomplete examinations due to poor tolerance

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study included patients with digestive diseases who were admitted to the First Affiliated Hospital of Sun Yat-sen University between July 2025 and August 2026.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The area under the ROC curve (AUC) to assess the performance of diagnostic model. | 6 months
  After baseline MR or CT scanning, patients were followed up.

CONTACTS AND LOCATIONS:
Overall Officials: Xuehua Li, Principal Investigator — Sun Yat-sen University First Affiliated Hospital Department of Radiology
Locations (1):
- XploreMET v3.0 system, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided